CLINICAL TRIAL: NCT02489318
Title: A Phase 3 Randomized, Placebo-controlled, Double-blind Study of Apalutamide Plus Androgen Deprivation Therapy (ADT) Versus ADT in Subjects With Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
Brief Title: A Study of Apalutamide (JNJ-56021927, ARN-509) Plus Androgen Deprivation Therapy (ADT) Versus ADT in Participants With mHSPC
Acronym: TITAN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR107614; 56021927PCR3002 (Other: Janssen Research & Development, LLC); 2015-000735-32 (EudraCT Number)
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; JNJ-56021927; Androgen Deprivation Therapy; ARN-509; Apalutamide; TITAN; Metastatic Hormone-sensitive Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Apalutamide plus ADT (Experimental): Participants will receive apalutamide 240 milligram (mg) (4X 60 mg tablets) with ADT.
  Interventions: Drug: Apalutamide; Drug: Androgen Deprivation Therapy (ADT)
- Placebo plus ADT (Experimental): Participants will receive matching Placebo with ADT.
  Interventions: Drug: Placebo; Drug: Androgen Deprivation Therapy (ADT)

INTERVENTIONS:
Drug: Apalutamide — Participants will receive apalutamide 240 mg (4 x 60 mg) tablets orally once daily in each 28 day treatment cycles.
  Other Names: JNJ-56021927; ARN-509
  Arms: Apalutamide plus ADT
Drug: Placebo — Participants will receive Placebo orally once daily in each 28 day treatment cycles.
  Arms: Placebo plus ADT
Drug: Androgen Deprivation Therapy (ADT) — All participants will receive and remain on a stable regimen of ADT (gonadotropin releasing hormone analog [GnRHa] or surgical castration). The choice of the GnRHa (agonist or antagonist) will be at discretion of the Investigator. Dosing (dose and frequency of administration) will be consistent with the prescribing information.

SUMMARY:
The purpose of this study is to determine if the addition of apalutamide to ADT provides superior efficacy in improving radiographic progression-free survival (rPFS) or overall survival (OS) for participants with mHSPC.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled, multinational, multicenter study of apalutamide in participants with mHSPC. The study consists of 4 Phases: Screening Phase (up to 28 days before randomization), Treatment Phase (28 day treatment cycles until disease progression or the occurrence of unacceptable treatment related toxicity), an End of Treatment Phase (until 30 days after the last dose of study drug), and then a Survival Follow up Phase. In the event of a positive study result and notification of unblinding at either of the interim analyses or at the final analysis, participants in the treatment Phase will have the opportunity to enroll in an Open-label Extension Phase, which will allow participants to receive active drug (apalutamide) for approximately 3 years. Participants who are receiving apalutamide in the Open-label Extension Phase may continue receiving apalutamide in the Long-term Extension (LTE) Phase if they will continue to derive benefit from treatment (based on investigator assessment). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate adenocarcinoma as confirmed by the investigator
* Metastatic disease documented by greater than or equal to (>=) 1 bone lesions on 99mTc bone scan. Participants with a single bone lesion must have confirmation of bone metastasis by computed tomography (CT) or magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) grade of 0 or 1
* Participants who received docetaxel treatment must meet the following criteria: a) Received a maximum of 6 cycles of docetaxel therapy for mHSPC; b) Received the last dose of docetaxel <=2 months prior to randomization; c) Maintained a response to docetaxel of stable disease or better, by investigator assessment of imaging and PSA, prior to randomization
* Other allowed prior treatment for mHSPC: a) Maximum of 1 course of radiation or surgical intervention; radiation therapy for metastatic lesions must be completed prior to randomization; b) Less than or equal to (<=) 6 months of ADT prior to randomization
* Allowed prior treatments for localized prostate cancer (all treatments must have been completed >= 1 year prior to randomization) a) <= 3 years total of ADT; b) All other forms of prior therapies including radiation therapy, prostatectomy,lymph node dissection, and systemic therapies

Exclusion Criteria:

* Pathological finding consistent with small cell, ductal or neuroendocrine carcinoma of the prostate
* Known brain metastases
* Lymph nodes as only sites of metastases
* Visceral (ie, liver or lung) metastases as only sites of metastases
* Other prior malignancy less than or equal to 5 years prior to randomization with the exception of squamous or basal cell skin carcinoma or non-invasive superficial bladder cancer
* Prior treatment with other next generation anti-androgens or other CYP17 inhibitors, immunotherapy or radiopharmaceutical agents for prostate cancer
* History of seizures or medications known to lower seizure threshold

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (222):
- United States (40):
  - Homewood, Alabama
  - Tucson, Arizona
  - San Bernardino, California
  - San Diego, California
  - Denver, Colorado
  - Norwalk, Connecticut
  - Fort Myers, Florida
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - Jeffersonville, Indiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - Lansing, Michigan
  - Troy, Michigan
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Brooklyn, New York
  - Poughkeepsie, New York
  - Syracuse, New York
  - The Bronx, New York
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Springfield, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Bryn Mawr, Pennsylvania
  - Lancaster, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Burien, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Argentina (12):
  - Berazategui
  - Buenos Aires
  - C.a.b.a.
  - Capital Federal
  - Ciudad Automoma Buenos Aires
  - Ciudad de Buenos Aires
  - Córdoba
  - La Plata
  - Pergamino
  - Rosario
  - San Miguel de Tucumán
  - San Salvador de Jujuy
- Australia (6):
  - Albury
  - Elizabeth Vale
  - Kogarah
  - Port Macquarie
  - South Brisbane
  - St Leonards
- Brazil (11):
  - Barretos
  - Florianópolis
  - Goiânia
  - Ijuí
  - Natal
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - Santo André
  - São Paulo
  - Sorocaba
- Canada (6):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Kingston, Ontario
  - Toronto, Ontario
  - Québec, Quebec
- China (12):
  - Beijing
  - Chengdu
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Suzhou
  - Wuhan
  - Wuxi
  - Xi'an
- Czechia (8):
  - Hradec Králove
  - Liberec
  - Nový Jicin
  - Olomouc
  - Opava
  - Pardubice
  - Prague
  - Zlín
- France (7):
  - Clermont-Ferrand
  - Montpellier
  - Nancy
  - Paris
  - Pierre-Bénite
  - Strasbourg
  - Suresnes
- Germany (10):
  - Bonn
  - Braunschweig
  - Eisleben Lutherstadt
  - Hamburg
  - Hanover
  - Leipzig
  - Lübeck
  - Nürtingen
  - Sindelfingen
  - Straubing
- Hungary (4):
  - Budapest
  - Győr
  - Pécs
  - Sopron
- Israel (7):
  - Beersheba
  - Haifa
  - Holon
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Zrifin
- Japan (14):
  - Chūōku
  - Hakata-Ku
  - Koshigaya
  - Matsuyama
  - Minamiku
  - Miyazaki
  - Nagano
  - Nagasaki
  - Osaka
  - Osaka Sayama Shi
  - Sakura
  - Sapporo
  - Yokohama
  - Yufu
- Mexico (7):
  - Durango
  - Guadalajara
  - León
  - Mexico City
  - México
  - Morelia
  - Zapopan
- Poland (10):
  - Bialystok
  - Bydgoszcz
  - Krakow
  - Kutno
  - Lodz
  - Lublin
  - Siedlce
  - Sochaczew
  - Warsaw
  - Wroclaw
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Târgu Mureş
- Russia (17):
  - Barnaul
  - Ivanovo
  - Moscow
  - Nizhny Novgorod
  - Obninsk
  - Omsk
  - Pyatigorsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Saransk
  - Sochi
  - Tambov
  - Tomsk
  - Tyumen
  - Ufa
  - Vologda
- South Korea (6):
  - Daegu
  - Daejeon
  - Goyang-si
  - Jeollanam-do
  - Seongnam-si
  - Seoul
- Spain (5):
  - Barcelona
  - Córdoba
  - Jerez de la Frontera
  - Madrid
  - Pamplona
- Sweden (7):
  - Gothenburg
  - Malmo
  - Örebro
  - Stockholm
  - Umeå
  - Uppsala
  - Vaxjo
- Turkey (Türkiye) (5):
  - Ankara
  - Edirne
  - Istanbul
  - Izmir
  - Mersin
- Ukraine (14):
  - Cherkasy
  - Dnipo
  - Dnipro
  - Ivano-Frankivsk
  - Khakhiv
  - Kharkiv
  - Khmelnytsky
  - Kyiv
  - Lviv
  - Odesa
  - Poltava
  - Uzhhorod
  - Vinnitsa
  - Zaporizhzhya
- United Kingdom (10):
  - Carlisle
  - Dundee
  - Glasgow
  - London
  - Newcastle upon Tyne
  - Oxford
  - Plymouth
  - Scunthorpe
  - Stockton-on-Tees
  - Wolverhampton

REFERENCES:
- [Derived] Karsh LI, Bevans KB, Saad F, Chung BH, Oudard S, Brookman-May SD, McCarthy SA, Smith MR, Chi KN, Small EJ, Agarwal N. Prostate-specific antigen and health-related quality of life in individuals with advanced prostate cancer treated with apalutamide: a plain language summary of the SPARTAN and TITAN studies. Future Oncol. 2024;20(35):2689-2698. doi: 10.1080/14796694.2024.2384257. Epub 2024 Aug 20. PMID 39163505
- [Derived] Merseburger AS, Agarwal N, Bjartell A, Uemura H, Soto AJ, Bhaumik A, Bohm J, Tran N, Krochmann N, Nematian-Samani M, Mundle SD, Brookman-May SD, Lopez-Gitlitz A, McCarthy SA, Chi K, Chowdhury S. Targeted Investigational Treatment Analysis of Novel Anti-androgen (TITAN) study: ultralow prostate-specific antigen decline with apalutamide plus androgen-deprivation therapy. BJU Int. 2024 Dec;134(6):982-991. doi: 10.1111/bju.16449. Epub 2024 Jun 28. PMID 38940282
- [Derived] Shen J, Chowdhury S, Agarwal N, Karsh LI, Oudard S, Gartrell BA, Feyerabend S, Saad F, Pieczonka CM, Chi KN, Brookman-May SD, Rooney B, Bhaumik A, McCarthy SA, Bevans KB, Mundle SD, Small EJ, Smith MR, Graff JN. Apalutamide efficacy, safety and wellbeing in older patients with advanced prostate cancer from Phase 3 randomised clinical studies TITAN and SPARTAN. Br J Cancer. 2024 Jan;130(1):73-81. doi: 10.1038/s41416-023-02492-8. Epub 2023 Nov 11. PMID 37951974
- [Derived] Merseburger AS, Agarwal N, Bhaumik A, Lefresne F, Karsh LI, Pereira de Santana Gomes AJ, Soto AJ, Given RW, Brookman-May SD, Mundle SD, McCarthy SA, Uemura H, Chowdhury S, Chi KN, Bjartell A. Apalutamide plus androgen deprivation therapy in clinical subgroups of patients with metastatic castration-sensitive prostate cancer: A subgroup analysis of the randomised clinical TITAN study. Eur J Cancer. 2023 Nov;193:113290. doi: 10.1016/j.ejca.2023.113290. Epub 2023 Aug 11. PMID 37708629
- [Derived] Agarwal N, McQuarrie K, Bjartell A, Chowdhury S, Pereira de Santana Gomes AJ, Chung BH, Ozguroglu M, Juarez Soto A, Merseburger AS, Uemura H, Ye D, Given R, Basch E, Miladinovic B, Lopez-Gitlitz A, Chi KN. Apalutamide plus Androgen Deprivation Therapy for Metastatic Castration-Sensitive Prostate Cancer: Analysis of Pain and Fatigue in the Phase 3 TITAN Study. J Urol. 2021 Oct;206(4):914-923. doi: 10.1097/JU.0000000000001841. Epub 2021 May 27. PMID 34039013
- [Derived] Chi KN, Chowdhury S, Bjartell A, Chung BH, Pereira de Santana Gomes AJ, Given R, Juarez A, Merseburger AS, Ozguroglu M, Uemura H, Ye D, Brookman-May S, Mundle SD, McCarthy SA, Larsen JS, Sun W, Bevans KB, Zhang K, Bandyopadhyay N, Agarwal N. Apalutamide in Patients With Metastatic Castration-Sensitive Prostate Cancer: Final Survival Analysis of the Randomized, Double-Blind, Phase III TITAN Study. J Clin Oncol. 2021 Jul 10;39(20):2294-2303. doi: 10.1200/JCO.20.03488. Epub 2021 Apr 29. PMID 33914595
- [Derived] Uemura H, Koroki Y, Iwaki Y, Imanaka K, Kambara T, Lopez-Gitlitz A, Smith A, Uemura H. Skin rash following Administration of Apalutamide in Japanese patients with Advanced Prostate Cancer: an integrated analysis of the phase 3 SPARTAN and TITAN studies and a phase 1 open-label study. BMC Urol. 2020 Sep 2;20(1):139. doi: 10.1186/s12894-020-00689-0. PMID 32878613
- [Derived] Agarwal N, McQuarrie K, Bjartell A, Chowdhury S, Pereira de Santana Gomes AJ, Chung BH, Ozguroglu M, Juarez Soto A, Merseburger AS, Uemura H, Ye D, Given R, Cella D, Basch E, Miladinovic B, Dearden L, Deprince K, Naini V, Lopez-Gitlitz A, Chi KN; TITAN investigators. Health-related quality of life after apalutamide treatment in patients with metastatic castration-sensitive prostate cancer (TITAN): a randomised, placebo-controlled, phase 3 study. Lancet Oncol. 2019 Nov;20(11):1518-1530. doi: 10.1016/S1470-2045(19)30620-5. Epub 2019 Sep 29. PMID 31578173
- [Derived] Chi KN, Agarwal N, Bjartell A, Chung BH, Pereira de Santana Gomes AJ, Given R, Juarez Soto A, Merseburger AS, Ozguroglu M, Uemura H, Ye D, Deprince K, Naini V, Li J, Cheng S, Yu MK, Zhang K, Larsen JS, McCarthy S, Chowdhury S; TITAN Investigators. Apalutamide for Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2019 Jul 4;381(1):13-24. doi: 10.1056/NEJMoa1903307. Epub 2019 May 31. PMID 31150574

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, 208 participants randomized to receive placebo+ADT were switched over to receive apalutamide+ADT after interim analysis and unblinding. Randomized treatment disposition has been reported in participant flow. Response/progression that occurred during a non-randomized switch-over to apalutamide+ADT were not counted towards efficacy outcome measures.
Groups:
- Placebo + Androgen Deprivation Therapy (ADT): Participants received matching placebo (4 tablets) orally once daily (qd) along with ADT (gonadotropin releasing hormone analog [GnRHa] or surgical castration) as standard of care therapy in each 28-day treatment cycle. The choice of the GnRHa (agonist or antagonist) was at discretion of the investigator. In the event of a positive result at interim or final analysis participants in treatment phase had opportunity to receive Apalutamide +ADT. Participants received treatment until radiographic progression or unequivocal clinical progression, unacceptable toxicity, or death.
- Apalutamide + ADT: Participants received JNJ-56021927 (apalutamide) 240 milligrams (mg) (4*60 mg tablets) orally qd along with ADT (gonadotropin releasing hormone analog [GnRHa] or surgical castration) as standard of care therapy in each 28-day treatment cycle. The choice of the GnRHa (agonist or antagonist) was at discretion of the investigator. Participants received treatment until radiographic progression or unequivocal clinical progression, unacceptable toxicity, or death.
Period: Randomized
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT
Started | 527 | 525
Completed | 527 | 524
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treated
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT
Started | 527 | 524
Completed | 208 (Participants crossed over from placebo to apalutamide after positive results at interim analysis.) | 0
Not Completed | 319 | 524
Not completed — Adverse Event | 19 | 62
Not completed — Death | 13 | 11
Not completed — Physician Decision | 4 | 6
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 37 | 36
Not completed — Other: Progressive Disease | 245 | 138
Not completed — Other | 0 | 2
Not completed — Ongoing | 0 | 267

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT | Total
Number analyzed (Participants) | 527 | 525 | 1052
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (8.42) | 68.9 (8.11) | 68.4 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 527 | 525 | 1052
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 6 | 17
  Asian | 112 | 119 | 231
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 365 | 354 | 719
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 30 | 35 | 65
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 20 | 17 | 37
  AUSTRALIA | 5 | 6 | 11
  BRAZIL | 38 | 54 | 92
  CANADA | 16 | 14 | 30
  CHINA | 46 | 48 | 94
  CZECH REPUBLIC | 12 | 19 | 31
  FRANCE | 8 | 8 | 16
  GERMANY | 10 | 7 | 17
  HUNGARY | 11 | 13 | 24
  ISRAEL | 8 | 6 | 14
  ITALY | 18 | 16 | 34
  JAPAN | 23 | 28 | 51
  MEXICO | 25 | 23 | 48
  POLAND | 12 | 7 | 19
  ROMANIA | 7 | 4 | 11
  RUSSIAN FEDERATION | 66 | 65 | 131
  SOUTH KOREA | 41 | 35 | 76
  SPAIN | 12 | 8 | 20
  SWEDEN | 8 | 8 | 16
  TURKEY | 22 | 28 | 50
  UKRAINE | 60 | 42 | 102
  UNITED KINGDOM | 16 | 20 | 36
  UNITED STATES | 43 | 49 | 92
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 11 | 6 | 17
  Asian | 112 | 119 | 231
  Black or African American | 9 | 10 | 19
  More than one race | 0 | 1 | 1
  Not Reported | 8 | 11 | 19
  Other | 22 | 24 | 46
  White | 365 | 354 | 719

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-free Survival (rPFS)
Description: rPFS as assessed by the investigator was defined as the duration from the date of randomization to the date of first documentation of radiographic progressive disease or death due to any cause, whichever occurred first. Radiographic progressive disease was defined as progression of soft tissue lesions measured by computed tomography (CT) or magnetic resonance imaging (MRI) as defined by modified Response evaluation criteria in solid tumors (RECIST) 1.1.
Time Frame: Up to 35 months
Population: Intent to treat (ITT) population included all randomized participants classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT
Number analyzed (Participants) | 527 | 525
months | 22.08 [18.46 to 32.92] | NA [NA to NA] — Here NA signifies that the median, lower limit and upper limit of confidence interval (CI) were not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Placebo + Androgen Deprivation Therapy (ADT) vs Apalutamide + ADT; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.484, 95% CI 2-sided [0.391 to 0.600]

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death from any cause.
Time Frame: Up to 57 months
Population: ITT population included all randomized participants classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT
Number analyzed (Participants) | 527 | 525
months | 52.17 [41.86 to NA] — Here NA signifies that the upper limit of CI was not estimable due to lesser number of events. | NA [NA to NA] — Here NA signifies that the median, lower limit and upper limit of CI were not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Placebo + Androgen Deprivation Therapy (ADT) vs Apalutamide + ADT; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.651, 95% CI 2-sided [0.534 to 0.793]

3. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy
Description: Time to initiation of cytotoxic chemotherapy was defined as the time from date of randomization to the date of initiation of cytotoxic chemotherapy for prostate cancer.
Time Frame: Up to 57 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT
Number analyzed (Participants) | 527 | 525
months | NA [NA to NA] — Here NA signifies that the median, lower limit and upper limit of CI were not estimable due to lesser number of events. | NA [NA to NA] — Here NA signifies that the median, lower limit and upper limit of CI were not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Placebo + Androgen Deprivation Therapy (ADT) vs Apalutamide + ADT; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.469, 95% CI 2-sided [0.350 to 0.630]

4. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was defined as the time from the date of randomization to the date of the first observation of pain progression. Pain progression was defined as an average increase by 2 points from baseline to greater than (>) 4 on the Brief Pain Inventory - Short Form (BPI-SF) worst pain intensity (item 3) with no decrease in opioids confirmed greater than equal to (>=) 3 weeks apart or initiation of chronic opioids, whichever occurred first. BPI-SF is a self-administered questionnaire developed to assess severity of pain and impact of pain on daily functions. Item 3 (worst pain intensity) asks participants to rate worst pain in prior 7-days on a 0-10 numeric rating scale, where "0" indicates "No pain" and "10" indicates "Pain as bad as you can imagine." A lower score is better.
Time Frame: Up to 57 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT
Number analyzed (Participants) | 527 | 525
months | NA [51.32 to NA] — Here NA signifies that the median and upper limit of CI were not estimable due to lesser number of events. | NA [NA to NA] — Here NA signifies that the median, lower limit and upper limit of CI were not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Placebo + Androgen Deprivation Therapy (ADT) vs Apalutamide + ADT; Test type: Superiority; p = 0.1966, Log Rank; Hazard Ratio (HR) = 0.868, 95% CI 2-sided [0.700 to 1.076]

5. Secondary Outcome: Time to Chronic Opioid Use
Description: Time to chronic opioid use was defined as the time from date of randomization to the first date of confirmed chronic opioid use. For participants entering the study without receiving opioids, chronic opioid use was defined as administration of opioid analgesics lasting for greater than or equal to (>=) 3 weeks for oral or >=7 days for non-oral formulations. For participants entering the study already receiving opioids, chronic opioid use was defined as a >=30 percent (%) increase in total daily dose of the opioid analgesics lasting for >= 3 weeks for oral or >= 7 days for non-oral formulation.
Time Frame: Up to 57 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT
Number analyzed (Participants) | 527 | 525
months | NA [51.32 to NA] — Here NA signifies that the median and upper limit of CI was not estimable due to lesser number of events. | NA [NA to NA] — Here NA signifies that the median, lower limit and upper limit of CI were not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Placebo + Androgen Deprivation Therapy (ADT) vs Apalutamide + ADT; Test type: Superiority; p = 0.1563, Log Rank; Hazard Ratio (HR) = 0.794, 95% CI 2-sided [0.576 to 1.094]

6. Secondary Outcome: Time to Skeletal-related Event (SRE)
Description: Time to SRE was defined as the time from the date of randomization to the date of the first observation of an SRE. A SRE was defined as the occurrence of either a pathological fracture, or spinal cord compression, or radiation to bone, or surgery to bone.
Time Frame: Up to 57 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Apalutamide + ADT
Number analyzed (Participants) | 527 | 525
months | NA [51.78 to NA] — Here NA signifies that the median and upper limit of CI were not estimable due to lesser number of events. . | NA [NA to NA] — Here NA signifies that the median, lower limit and upper limit of CI were not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Placebo + Androgen Deprivation Therapy (ADT) vs Apalutamide + ADT; Test type: Superiority; p = 0.3608, Log Rank; Hazard Ratio (HR) = 0.857, 95% CI 2-sided [0.615 to 1.194]

ADVERSE EVENTS:
Time Frame: Up to 57 months
Description: Safety Analysis set included all participants who received at least 1 dose of randomized study drug. Crossover participants were counted twice (in Placebo + ADT arm and in Placebo + ADT to Apalutamide + ADT arm) for safety analysis. For crossover participants, adverse events after initiation of crossover treatment were summarized separately in Placebo + ADT to Apalutamide + ADT arm. However, adverse events occurred before crossover treatment were summarized in Placebo + ADT arm.
Groups:
- Placebo + ADT to Apalutamide + ADT: After interim analysis and unblinding, participants receiving placebo +ADT crossed over to receive 240 mg apalutamide orally qd along with ADT in open-label extension phase.
Arm/Group | Placebo + Androgen Deprivation Therapy (ADT) | Placebo + ADT to Apalutamide + ADT | Apalutamide + ADT
All-Cause Mortality (participants affected / at risk) | 35/527 | 10/208 | 31/524
Serious Adverse Events (participants affected / at risk) | 115/527 | 29/208 | 153/524
Other Adverse Events (participants affected / at risk) | 485/527 | 153/208 | 494/524
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Androgen Deprivation Therapy (ADT) (N=527) | Placebo + ADT to Apalutamide + ADT (N=208) | Apalutamide + ADT (N=524)
Anaemia (Blood and lymphatic system disorders) | 6 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 3
Angina Pectoris (Cardiac disorders) | 2 | 0 | 3
Angina Unstable (Cardiac disorders) | 1 | 0 | 0
Aortic Valve Disease Mixed (Cardiac disorders) | 0 | 0 | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 2
Atrioventricular Block Complete (Cardiac disorders) | 0 | 0 | 1
Cardiac Amyloidosis (Cardiac disorders) | 1 | 0 | 0
Cardiac Disorder (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 2
Cor Pulmonale Chronic (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Stenosis (Cardiac disorders) | 0 | 0 | 3
Mitral Valve Disease (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 8
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1
Sinoatrial Block (Cardiac disorders) | 0 | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 0 | 0 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 1
Vertigo Positional (Ear and labyrinth disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Open Angle Glaucoma (Eye disorders) | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 2
Anal Fistula (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhagic Erosive Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 3
Large Intestinal Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2
Terminal Ileitis (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 2
Exercise Tolerance Decreased (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0
Gait Disturbance (General disorders) | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 2 | 0
Oedema (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Performance Status Decreased (General disorders) | 0 | 0 | 1
Peripheral Swelling (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholangiolitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal Abscess (Infections and infestations) | 1 | 0 | 0
Abscess Jaw (Infections and infestations) | 1 | 0 | 0
Abscess Oral (Infections and infestations) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 3
Cellulitis (Infections and infestations) | 2 | 0 | 0
Cholecystitis Infective (Infections and infestations) | 0 | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1
Fournier's Gangrene (Infections and infestations) | 1 | 0 | 0
Infected Lymphocele (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Kidney Infection (Infections and infestations) | 1 | 0 | 0
Klebsiella Infection (Infections and infestations) | 1 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Muscle Abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 3 | 10
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 2 | 2 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 5
Urosepsis (Infections and infestations) | 1 | 0 | 5
Viral Infection (Infections and infestations) | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brain Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Comminuted Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skull Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4
Subarachnoid Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
International Normalised Ratio Increased (Investigations) | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 3
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Adrenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Burkitt's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung Carcinoma Cell Type Unspecified Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Respiratory Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cauda Equina Syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 3 | 4
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 1
Diplegia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1 | 1
Iiird Nerve Paresis (Nervous system disorders) | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 6 | 0 | 2
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1 | 2
Device Malfunction (Product Issues) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 2
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 3
Bladder Perforation (Renal and urinary disorders) | 1 | 0 | 0
Bladder Tamponade (Renal and urinary disorders) | 1 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 1 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 3
Haematuria (Renal and urinary disorders) | 3 | 1 | 10
Hydronephrosis (Renal and urinary disorders) | 4 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal Disorder (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 2
Ureterolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 2 | 0 | 0
Urinary Bladder Haematoma (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 9 | 0 | 4
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 3
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 | 1 | 2
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Paranasal Cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 3
Venous Stenosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Androgen Deprivation Therapy (ADT) (N=527) | Placebo + ADT to Apalutamide + ADT (N=208) | Apalutamide + ADT (N=524)
Anaemia (Blood and lymphatic system disorders) | 71 | 13 | 68
Leukopenia (Blood and lymphatic system disorders) | 21 | 8 | 29
Neutropenia (Blood and lymphatic system disorders) | 15 | 2 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 6 | 12
Hypothyroidism (Endocrine disorders) | 5 | 5 | 23
Abdominal Pain (Gastrointestinal disorders) | 22 | 3 | 17
Abdominal Pain Upper (Gastrointestinal disorders) | 13 | 2 | 17
Constipation (Gastrointestinal disorders) | 57 | 6 | 58
Diarrhoea (Gastrointestinal disorders) | 35 | 11 | 56
Dyspepsia (Gastrointestinal disorders) | 10 | 2 | 12
Nausea (Gastrointestinal disorders) | 44 | 12 | 41
Toothache (Gastrointestinal disorders) | 11 | 1 | 10
Vomiting (Gastrointestinal disorders) | 23 | 3 | 22
Asthenia (General disorders) | 45 | 8 | 40
Fatigue (General disorders) | 87 | 15 | 107
Influenza Like Illness (General disorders) | 17 | 3 | 16
Oedema Peripheral (General disorders) | 41 | 4 | 32
Pyrexia (General disorders) | 16 | 4 | 15
Bronchitis (Infections and infestations) | 12 | 1 | 18
Conjunctivitis (Infections and infestations) | 5 | 2 | 13
Herpes Zoster (Infections and infestations) | 11 | 0 | 10
Influenza (Infections and infestations) | 23 | 5 | 21
Nasopharyngitis (Infections and infestations) | 47 | 6 | 44
Pneumonia (Infections and infestations) | 14 | 4 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 29 | 6 | 40
Urinary Tract Infection (Infections and infestations) | 22 | 4 | 28
Contusion (Injury, poisoning and procedural complications) | 11 | 4 | 11
Fall (Injury, poisoning and procedural complications) | 36 | 8 | 47
Rib Fracture (Injury, poisoning and procedural complications) | 14 | 1 | 14
Alanine Aminotransferase Increased (Investigations) | 42 | 4 | 25
Aspartate Aminotransferase Increased (Investigations) | 43 | 5 | 18
Blood Alkaline Phosphatase Increased (Investigations) | 32 | 3 | 18
Blood Lactate Dehydrogenase Increased (Investigations) | 17 | 0 | 9
Blood Thyroid Stimulating Hormone Increased (Investigations) | 2 | 3 | 16
Weight Decreased (Investigations) | 29 | 9 | 43
Weight Increased (Investigations) | 92 | 7 | 55
Decreased Appetite (Metabolism and nutrition disorders) | 27 | 11 | 32
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 | 7 | 34
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 1 | 18
Hyperkalaemia (Metabolism and nutrition disorders) | 27 | 16 | 47
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13 | 5 | 22
Hyponatraemia (Metabolism and nutrition disorders) | 16 | 2 | 7
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 82 | 15 | 101
Back Pain (Musculoskeletal and connective tissue disorders) | 108 | 11 | 106
Bone Pain (Musculoskeletal and connective tissue disorders) | 53 | 0 | 39
Groin Pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 11
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 10 | 2 | 21
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 12 | 2 | 18
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 15 | 2 | 21
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 41 | 5 | 39
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 2 | 10
Osteoporosis (Musculoskeletal and connective tissue disorders) | 7 | 0 | 16
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 67 | 8 | 69
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 5 | 0 | 11
Spinal Pain (Musculoskeletal and connective tissue disorders) | 12 | 3 | 13
Dizziness (Nervous system disorders) | 35 | 7 | 24
Dysgeusia (Nervous system disorders) | 2 | 2 | 13
Headache (Nervous system disorders) | 31 | 12 | 44
Hypoaesthesia (Nervous system disorders) | 12 | 1 | 9
Paraesthesia (Nervous system disorders) | 15 | 0 | 11
Anxiety (Psychiatric disorders) | 6 | 1 | 11
Insomnia (Psychiatric disorders) | 33 | 5 | 28
Dysuria (Renal and urinary disorders) | 30 | 3 | 35
Haematuria (Renal and urinary disorders) | 14 | 3 | 21
Nocturia (Renal and urinary disorders) | 15 | 1 | 16
Pollakiuria (Renal and urinary disorders) | 19 | 5 | 21
Urinary Incontinence (Renal and urinary disorders) | 8 | 0 | 14
Urinary Retention (Renal and urinary disorders) | 14 | 0 | 13
Pelvic Pain (Reproductive system and breast disorders) | 14 | 1 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 4 | 40
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 13
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 13
Dry Skin (Skin and subcutaneous tissue disorders) | 8 | 2 | 18
Eczema (Skin and subcutaneous tissue disorders) | 7 | 4 | 12
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3 | 14
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 | 1 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 13 | 58
Rash (Skin and subcutaneous tissue disorders) | 23 | 26 | 106
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 6 | 17
Hot Flush (Vascular disorders) | 87 | 3 | 121
Hypertension (Vascular disorders) | 84 | 13 | 100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02489318/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT02489318/SAP_001.pdf